CLINICAL TRIAL: NCT00006161
Title: Decompression Intervention of Variceal Rebleeding Trial
Brief Title: Decompression Intervention of Variceal Rebleeding Trial (DIVERT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: DIVERT (completed); DK50680-02; NCT00004469 (obsolete NCT alias)
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Esophageal and Gastric Varices; Liver Cirrhosis
Keywords: TIPS; DSRS; Varices; Variceal bleeding; Splenorenal Shunt; Transjugular Intrahepatic Portosystemic Shunt; Cirrhosis; Portal hypertension; Liver disease
MeSH Terms: conditions — Esophageal and Gastric Varices; Liver Cirrhosis; Varicose Veins; Fibrosis; Hypertension, Portal; Liver Diseases | interventions — Portasystemic Shunt, Transjugular Intrahepatic

INTERVENTIONS:
Procedure: Transjugular Intrahepatic Portosystemic Shunt (TIPS)
Procedure: Distal Splenorenal Shunt

SUMMARY:
The Decompression Intervention of Variceal Rebleeding Trial (DIVERT) is a multi-center prospective randomized clinical trial comparing the radiologic procedure of transjugular intrahepatic portal-systemic shunt (TIPS) with the surgical procedure of distal splenorenal shunt (DSRS) for variceal bleeding in patients with Child's Class A and B cirrhosis.

This is recognized nationally and internationally as the study that will answer the question as to which of these is the best treatment for decompression of varices in patients who have failed endoscopic and pharmacologic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Variceal bleeding secondary to cirrhosis and portal hypertension
* Child's Class A or B cirrhosis of any etiology
* Patients who have failed endoscopic therapy (sclerotherapy or banding) of varices; or patients who are not candidates for endoscopic therapy

Exclusion Criteria:

* Prior shunt procedure
* Portal vein thrombosis
* Polycystic liver disease
* Intractable ascites
* Prior organ transplant
* Any medical intractable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 1996-12; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Henderson, M.D., Principal Investigator — The Cleveland Clinic; Thomas D. Boyer, M.D., Principal Investigator — Emory University; Lennox Jeffers, M.D., Principal Investigator — University of Miami; Enrique Molina, M.D., Principal Investigator — University of Miami; Layton F. Rikkers, M.D., Principal Investigator — University of Wisconsin, Madison; Kareem Abu-Elmagd, M.D., Principal Investigator — University of Pittsburgh Medical Center; Amrik Shah, Sc.D., Principal Investigator — Cleveland Clinic Foundation - Data Coordinating Center
Locations (5):
- United States (5):
  - University of Miami School of Medicine, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Boyer TD, Henderson JM, Heerey AM, Arrigain S, Konig V, Connor J, Abu-Elmagd K, Galloway J, Rikkers LF, Jeffers L; DIVERT Study Group. Cost of preventing variceal rebleeding with transjugular intrahepatic portal systemic shunt and distal splenorenal shunt. J Hepatol. 2008 Mar;48(3):407-14. doi: 10.1016/j.jhep.2007.08.014. Epub 2007 Oct 23. PMID 18045724